CLINICAL TRIAL: NCT02495324
Title: A Randomized, Double-blind, Active Control, 3-parallel Group, Forced Titration, Multicenter, Phase IV Study to Evaluate the Efficacy and Safety of Fimasartan Versus Valsartan Monotherapy in Patients With Mild to Moderate Essential Hypertension
Brief Title: Fimasartan Achieving SBP Target (FAST) Study
Acronym: FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BR-FVO-CT-401
Record Dates: First submitted 2015-07-07; First posted 2015-07-13 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Essential,Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Valsartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fimasartan (Experimental): Placebo daily for 2 weeks and Fimasartan 60mg daily for 2 weeks and 120mg daily for 4 weeks
  Interventions: Drug: Placebo; Drug: Fimasartan
- Valsartan (Active Comparator): Placebo daily for 2 weeks and Valsartan 80mg daily for 2 weeks and 160mg daily for 4 weeks
  Interventions: Drug: Placebo; Drug: Valsartan
- Olmesartan medoxomil (Other): Reference group. Placebo daily for 2 weeks and Olmesartan 10mg daily for 2 weeks and 20mg daily for 4 weeks
  Interventions: Drug: Placebo; Drug: Olmesartan medoxomil

INTERVENTIONS:
Drug: Placebo — 2 weeks of placebo PO daily
Drug: Fimasartan — 60mg 1 tab PO daily for 2 weeks and 120mg 1 tab PO daily for 4 weeks
  Other Names: Kanarb Tab
  Arms: Fimasartan
Drug: Valsartan — 80mg 1 tab PO daily for 2 weeks and 160mg 1 tab PO daily for 4 weeks
  Other Names: Diovan Tab
  Arms: Valsartan
Drug: Olmesartan medoxomil — 10mg 1 tab PO daily for 2 weeks and 20mg 1 tab PO daily for 4 weeks
  Other Names: Olmetec Tab
  Arms: Olmesartan medoxomil

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Fimasartan compared to Valsartan and Olmesartan(reference group) in patients with mild to moderate essential hypertension. Patients have 2 weeks of placebo run-in and wash out period, 2 weeks of taking required dose and 4 weeks of taking double dose.

DETAILED DESCRIPTION:
A randomized, double-blind, active control, 3-parallel group comparison clinical study to evaluate the anti-hypertensive efficacy and safety of Fimasartan in patients with mild to moderate hypertension. Approximately 360 patients will be enrolled in 8 centers in South Korea. This study has planned 6 visits during 8 weeks.(2 weeks of placebo run-in and wash out, 2 weeks of treatment and 4 weeks of forced titration) All of the subjects who agreed to participate in this study and gave written informed consent voluntarily are assessed the inclusion and exclusion criteria and receive the investigational product(placebo) at screening visit. During more than 14 days of placebo run-in and wash out period, subjects have to stop the previous anti-hypertensive drug. After placebo run-in and wash out period, Subjects are assessed the final eligibility and started measuring ambulatory blood pressure for 24 hours. Subjects who determined to be appropriate for this study are allocated to experimental group(Fimasartan 60mg) or control group(Valsartan 80mg) or Reference group(Olmesartan 10mg) randomly at ratio 3:3:1.Subjects take their investigational products daily for 2 weeks and double dose for 4 weeks. The placebo period will be single-blinded and the treatment allocation in this study will be double-blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily signed informed consent for participating in this clinical trial
2. Male and female between 19 and 70 years old
3. Subjects whose mean sitting SBP(siSBP) of 3 measurements is above 140mmHg at visit 2 with mild to moderate essential hypertension (Subjects who have not taken anti-hypertensive drugs within 3 months should have mean siSBP above 140mmHg at visit 1)
4. Subject who can understand the trial procedures and be willing to cooperate the trial

Exclusion Criteria:

1. Severe hypertension patients with mean siSBP ≥ 180mmHg or siDBP ≥110mmHg at the assessment of Screening visit(Visit1) and Baseline visit (Visit2).
2. Patients whose difference between maximum and minimum among 3 times of blood pressure measurement is over 20mmHg(siSBP) or 10mmHg(siDBP) at visit1 and visit2.
3. Patients whose medication compliance is under 70% at visit 2.
4. Secondary hypertension patients, but not limited to the following diseases (example: renovascular disease, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromocytoma, polycystic kidney disease, etc).
5. Patients who have postural hypotension with manifestation.
6. Subjects with severe insulin-dependent Diabetes Mellitus(DM) or uncontrolled DM(HbA1c > 9% at screening visit, modified dosage of an oral hypoglycemic agent within 12 weeks prior to screening visit, or currently use of active insulin treatment).
7. History of malignant tumor including leukemia and lymphoma in the past 5 years.
8. Subjects with chronic inflammatory disease requiring an chronic anti-inflammatory therapy, past or current medical history with wasting disease, autoimmune diseases (e.g. rheumatoid arthritis, systemic lupus erythematosus) or connective tissue disease.
9. Medical history with hypersensitivity to angiotensin II antagonist.
10. Clinically significant renal and liver disorders such as dialysis, cirrhosis, biliary obstruction, cholestasis and liver failure. Patients who have below abnormality in the laboratory results at screening visit.

    * Creatinine clearance(Cockroft-Gault)<30mL/min
    * ALT, AST ≥ 2 times upper normal limit
    * Clinically significant hypokalemia(K<3.5mmol/L) or hyperkalemia(K>5.5mmol/L)
11. Subjects have history of any of the followings within the past 6 months or determined clinically significant by investigators.

    * Severe heart disease (Heart failure New York Heart Association(NYHA) class 3 and 4), ischemic heart disease (angina pectoris, myocardial infarction), peripheral vascular disease, percutaneous transluminal coronary angioplasty or coronary artery bypass graft.
    * Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve stenosis, or mitral valve stenosis.
    * Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or any other clinical significant arrhythmia.
    * Severe cerebrovascular disorder(e.g.stroke, cerebral infarction or cerebral hemorrhage)
12. Subjects with known moderate or malignant retinosis in the past 6 months (e.g. retinal hemorrhage, visual disturbance or retinal microaneurysm)
13. Subjects with history of abusing drugs or alcohol within the past 2 years.
14. Pregnant women or lactating female.
15. Subjects with following surgical and internal disease that may affect absorption, distribution, metabolism or excretion of drugs and have conditions which include the following (but are not limited to): history of major gastrointestinal surgeries including gastrectomy, gastro-enterostomy or bowel resection, gastrointestinal bypass graft and stabling; current active gastritis, gastrointestinal and rectal bleeding, presence of active inflammatory bowel syndrome within the past 12 months.
16. Subjects with shock, depletion of body fluid or sodium ion not able to correct.
17. Subjects with hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
18. Medical history with clinically significant hypersensitivity to any components or other drugs on the investigational product or additives(yellow4 and yellow 5).
19. Subjects planning pregnancy or childbearing potential who are not using effective contraceptive methods.
20. Subjects who are participating in another trial or took other investigational product within 12 weeks prior to screening visit.
21. Subjects with other reasons not specified above and ineligible to participate in this clinical trial at discretion of study investigators.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change of sitting SBP from baseline after taking investigational products for 6 weeks. | 6 weeks from baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: KI-BAE SEUNG, Ph.D, Study Chair — Cardiovascular center, Seoul St.Mary's Hospital, The Catholic University of Korea
Locations (8):
- South Korea (8):
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, Banpo-dong, Seocho-gu
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Incheon, Bupyeong-gu
  - The Catholic University of Korea, St. Paul's Hospital, Seoul, Dongdaemun-gu
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea, St.Vincent's Hospital., Suwon, Gyeonggi-do
  - The Catholic University of Korea,Uijeongbu St.Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon, Jung-gu/Daeheung-ro
  - The Catholic University of Korea,Yeouido St.Mary's Hospital, Seoul, Yeongdeungpo-gu

REFERENCES:
- [Derived] Chung WB, Ihm SH, Jang SW, Her SH, Park CS, Lee JM, Chang K, Jeon DS, Yoo KD, Seung KB. Effect of Fimasartan versus Valsartan and Olmesartan on Office and Ambulatory Blood Pressure in Korean Patients with Mild-to-Moderate Essential Hypertension: A Randomized, Double-Blind, Active Control, Three-Parallel Group, Forced Titration, Multicenter, Phase IV Study (Fimasartan Achieving Systolic Blood Pressure Target (FAST) Study). Drug Des Devel Ther. 2020 Jan 23;14:347-360. doi: 10.2147/DDDT.S231293. eCollection 2020. PMID 32158190